CLINICAL TRIAL: NCT05773963
Title: A Post-market Study to Evaluate the Effects of Sodium Hyaluronate Based Eye Drops in Patients Affected by Dry Eye Disease.
Acronym: M-DED-2020
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Montefarmaco OTC SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M-DED-2020
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Opthalomology/Dry Eye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At V0, as per clinical practice, only 1 of the IPs products can be assigned to the enrolled subject (Other): At V0, as per clinical practice, only 1 of the IPs products can be assigned to the enrolled subject
  Interventions: Device: Irilens; Iridina; Afomill Lubricating Eye Drops

INTERVENTIONS:
Device: Irilens; Iridina; Afomill Lubricating Eye Drops — * Irilens (with 0.4% HA as key ingredient);
  * Iridina (with 0.4% HA as key ingredient);
  * Afomill Lubricating Eye Drops (with 0.2% HA as key ingredient and distilled water of Chamomile).

SUMMARY:
Dry eye disease (DED), also called keratoconjunctivitis sicca, is a multifactorial disease of the ocular surface characterized by loss of homeostasis of the tear film and accompanied by symptoms such as ocular discomfort and visual disturbance. The reported prevalence of DED estimates vary widely, from 5% to 33%, which may reflect both differing populations and inconsistent diagnostic criteria. Patients with moderate-to-severe DED may experience a reduced quality of life due to ocular pain, difficulty in performing daily activities, and depression. First-line therapy for treating dry eye consists of over the counter (OTC) artificial tear drops, gels, ointments, or lubricants.

Sodium hyaluronate (commonly referred to as hyaluronic acid or HA) is a naturally occurring polymer and is ubiquitous throughout the interstitial cellular space in humans. It helps retain moisture in different types of tissue throughout the human body and aids lubrication between layers of tissue to eliminate friction - thus making it an ideal physiological tear film substitute.

As a result of its coiled structure and large hydrophilic domains, HA attracts and retains a large amount of water, and therefore possesses the ability to retard water evaporation. Following instillation, HA-based solutions effectively moisturize the eye surface and prolong the beneficial wetting effect over time.

Hyaluronic acid does not alter the normal surface of the eye like other types of tear substitutes. It closely mimics the properties of a normal, healthy tear film, with a longer retention time on the corneal surface than a cellulose-based tear substitute.

HA gels have also been used successfully in ophthalmic surgery for many years. As a result of their unique physical and chemical properties, HA solutions are similar to natural tears. For that reason, they are widely used in ophthalmology as lubricant eye drops for the treatment of sensations of ocular dryness.

For these reasons, an interventional, confirmative, post marketing clinical follow-up (PMCF) study was planned to evaluate the performance and safety of HA-based ophthalmic solutions (i.e. Irilens; Iridina; Afomill Lubricating Eye Drops) used to relieve dry eyes symptoms.

The objectives of this PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of three investigational products (IPs) containing HA as key ingredient.

The IPs are on the market with the following brand names:

* Irilens;
* Iridina;
* Afomill Lubricating Eye Drops.

Primary

• To evaluate the performance of IPs used as intended to relieve dry eye symptoms.

Secondary

* To evaluate the efficacy of IPs used as intended to relieve symptoms of DED.
* To evaluate the safety and tolerability of the IPs.
* To evaluate the patient satisfaction of the IPs.

DETAILED DESCRIPTION:
Study Rationale: Dry eye disease (DED), also called keratoconjunctivitis sicca, is a multifactorial disease of the ocular surface characterized by loss of homeostasis of the tear film and accompanied by symptoms such as ocular discomfort and visual disturbance. The reported prevalence of DED estimates vary widely, from 5% to 33%, which may reflect both differing populations and inconsistent diagnostic criteria. Patients with moderate-to-severe DED may experience a reduced quality of life due to ocular pain, difficulty in performing daily activities, and depression. First-line therapy for treating dry eye consists of over the counter (OTC) artificial tear drops, gels, ointments, or lubricants.

Sodium hyaluronate (commonly referred to as hyaluronic acid or HA) is a naturally occurring polymer and is ubiquitous throughout the interstitial cellular space in humans. It helps retain moisture in different types of tissue throughout the human body and aids lubrication between layers of tissue to eliminate friction - thus making it an ideal physiological tear film substitute.

As a result of its coiled structure and large hydrophilic domains, HA attracts and retains a large amount of water, and therefore possesses the ability to retard water evaporation. Following instillation, HA-based solutions effectively moisturize the eye surface and prolong the beneficial wetting effect over time.

Hyaluronic acid does not alter the normal surface of the eye like other types of tear substitutes. It closely mimics the properties of a normal, healthy tear film, with a longer retention time on the corneal surface than a cellulose-based tear substitute.

HA gels have also been used successfully in ophthalmic surgery for many years. As a result of their unique physical and chemical properties, HA solutions are similar to natural tears. For that reason, they are widely used in ophthalmology as lubricant eye drops for the treatment of sensations of ocular dryness.

For these reasons, an interventional, confirmative, post marketing clinical follow-up (PMCF) study was planned to evaluate the performance and safety of HA-based ophthalmic solutions (i.e. Irilens; Iridina; Afomill Lubricating Eye Drops) used to relieve dry eyes symptoms.

Study Objective: The objectives of this PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of three investigational products (IPs) containing HA as key ingredient.

The IPs are on the market with the following brand names:

* Irilens;
* Iridina;
* Afomill Lubricating Eye Drops.

Primary • To evaluate the performance of IPs used as intended to relieve dry eye symptoms.

Secondary

* To evaluate the efficacy of IPs used as intended to relieve symptoms of DED.
* To evaluate the safety and tolerability of the IPs.
* To evaluate the patient satisfaction of the IPs.

Methodology: Potential candidates, that according the investigator judgment could be treated with one of IPs, will be identified, with the assessment of their eligibility criteria. Each subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), as per clinical practice, only one of the below reported IPs products can be assigned to the enrolled subject, depending on investigator clinical evaluation and decision:

* Irilens;
* Iridina;
* Afomill Lubricating Eye Drops.

The patient will perform 2 on site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

Data coming from additional assessments (e.g. blood tests), if done per clinical practice to perform DED diagnosis and evaluations, might be collected and used.

Number of subjects Planned: About 90 patients in total. Treatment duration: After baseline visit and IP dispensing, the treatment duration (according to the Investigation Product IFU) will be prolonged until the V2 (EOS visit; 25+ 5 days).

Safety Analysis Set (SAS): The "Safety Analysis Set" (SAS): this set included all enrolled patients who took at least one dose of IP.

Full Analysis Set (FAS): The "Full Analysis Set" (FAS): this set included all enrolled patients who took at least one dose of IP, and with a baseline and at least one post-baseline performance assessment.

Per protocol (PP): The "Per-Protocol" (PP) set: would include all the FAS patients who (a) met all inclusion/exclusion criteria liable to affect the performance assessment, (b) did not present serious deviations of the protocol that may affect efficacy.

I

IPs medical devices:

* Irilens (with 0.4% HA as key ingredient);
* Iridina (with 0.4% HA as key ingredient);
* Afomill Lubricating Eye Drops (with 0.2% HA as key ingredient and distilled water of Chamomile).

They are ophthalmic solutions with pH, isotonicity and osmolarity compatible with eye tissue and tear fluid.

Irilens, Iridina and Afomill Lubricating Eye Drops are suitable in the treatment of dry eyes symptomatology due to use of contact lenses, environmental reasons, excessive hours of study or computer work. Irilens and Iridina are suitable also after eye surgery.

Dose/dosage: All IPs are available as 10 ml multi-dose bottles. Irilens contains sodium chlorite as vanishing preservative. Iridina is a preservative-free ophthalmic solution. Afomill Lubricating Eye Drops contains Phmb 0.0002% as preservative.

Irilens is also available as preservative-free 0.5 ml mono-dose vials. The IP dosage for each individual case will be defined according to investigator judgment.

Administration:

The application of IP on eye surface should be performed in accordance to the indication for use.

According to the Investigator judgement, based on the subject clinical conditions and the indications reported on the IFU, one of the investigational products can be assigned to the subject to be enrolled in the trial.

The first administration and the intervals at which the treatment should be repeated, to be done as per investigator judgment and according the IFU, depend on various factors regarding the physiology of the patients (e.g. type of eye-tear film, anatomy, age), their lifestyle (e.g. use of computer, wearing of contact lenses).

Primary efficacy endpoint

• To evaluate the performance of IPs to relieve symptoms of dry eye, the Shirmer I test (ST) might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.

Secondary efficacy endpoints

* To assess the efficacy of IPs used as intended to relieve symptoms of dry eye, the difference of "Ocular surface index" (OSDI) Questionnaire between baseline (V0) and end of study visit (EOS/V2) will be evaluated stratified by study IPs.
* To assess the efficacy of IPs used as intended to relieve symptoms of dry eye, the Tear breakup time (TBUT) test might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.
* To evaluate the safety and tolerability of the IPs a Visual Analogue Scale (VAS) will be used.
* The patient satisfaction will be evaluated with a 5-points Likert Scale.

Safety:

Safety will be monitored through eye examination and adverse events including assessment of relationship to the IP.

Time-points for efficacy and safety: Baseline (V0) and follow up visit(s) performed.

Statistical methods:

Supposing a minimum difference of 20% (equals to 1 mm of difference) between after treatment and at baseline visit in terms of mean ST value, with a standard deviation (SD) equal to 1.7 mm, a correlation between baseline and end of treatment of 50%, and a type I error of 5%, 25 patients are sufficient to reach a statistical power greater than 80% for each IPs.

Moreover, planning to enroll a total of 30 patients would allow for a 15% drop-out rate.

Considering all IPs included, 90 patients should be enrolled in the study. In general, all the variables will be descriptively analyzed by treatment groups and visit (mean, median, standard deviation, minimum and maximum for continuous variables after normality check of distribution with Kolmogorov-Smirnov test, frequency distribution for categorical variables). All the analysis will be detailed in the Statistical Analysis Plan (SAP) which will be finalized in Version 1.0 before the Data Base Lock (DBL).

In details, the safety data will include (at least) physical examinations, laboratory data and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* M & F Aged ≥ 18 years at the time of the signature of ICF;
* Patients with ocular symptoms such as burning, itching, and foreign body sensation due to environmental factors, life habits, contact lenses wearing
* Diagnosis of mild-severe dry eye (OSDI score >8).
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions;
* Retinal pathology;
* Other type of ophthalmic neuropathy;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases);
* Known hypersensitivity or allergy to IP components;
* Eye surgery during the previous 3 months (e.g. LASIK, cataract surgery)
* Presence of any relevant severe organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant in Investigator's opinion;
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of Investigational Products to relieve symptoms of dry eye. The performance will be evaluated by Shirmer I test at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 25
  To evaluate the performance of IPs to relieve symptoms of dry eye, the Shirmer I test (ST) might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.

SECONDARY OUTCOMES:
Efficacy of Investigational Products used as intended to relieve symptoms of dry eye. The Efficacy will be evaluated by Questionnaire at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 25
  To assess the efficacy of IPs used as intended to relieve symptoms of dry eye, the difference of "Ocular surface index" (OSDI) Questionnaire between baseline (V0) and end of study visit (EOS/V2) will be evaluated stratified by study IPs.
To assess the efficacy of Investigational Products used as intended to relieve symptoms of dry eye. The efficacy will be evaluated by Tear breakup time test at baseline (V0) and end of study visit (change will be assessed) | Day 0 (baseline visit the IP will be dispensed) and Day 25
  To assess the efficacy of IPs used as intended to relieve symptoms of dry eye, the Tear breakup time (TBUT) test might be completed at baseline (V0) and end of study visit (EOS/V2). The evaluation will be performed stratified by study IPs.
Evaluation of the safety and tolerability of the Investigational Products by Visual Analogue Scale at the end of study visit | Day 25
  To evaluate the safety and tolerability of the IPs a Visual Analogue Scale (VAS) will be used.
The patient satisfaction will be evaluated with a 5-points Likert Scale at the end of study visit | Day 25
  The patient satisfaction will be evaluated with a 5-points Likert Scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Istituto Auxologico Italiano, Milan
  - Ospedale Felice Liotti Pontedera, Pisa